CLINICAL TRIAL: NCT06803563
Title: Effects of Physical Exercise and Motor Activity on Sleep Disorders in Post-Mastectomy Pain Syndrome
Brief Title: Physical Exercise, Motor Activity on Sleep Disorders in Post-Mastectomy Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Gioacchino Calapai (Other)
Responsible Party: Sponsor-Investigator, Gioacchino Calapai, Professor, Azienda Ospedaliera Universitaria Policlinico "G. Martino"
Organization: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Other Study IDs: BCMASD
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain Syndrome
Keywords: Chronic pain; post mastectomy; sleep disorders; physical activity; haematological markers
MeSH Terms: conditions — Chronic Pain; Sleep Wake Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pain is an unpleasant sensation common to all those who undergo surgery. Several studies indicate that 40-60% of patients experience the post-operative experience and can be caused by both internal and external stimuli. Chronic post mastectomy pain is a condition characterized by pain in the anterior chest, armpit, and/or upper arm, usually ipsilateral to surgery, which begins after mastectomy or quadrantectomy and persists for longer three months after surgery. It can become chronic in a broad spectrum of conditions. Psychosocial factors such as anxiety and sleep disturbance are being revealed as crucial contributors to individual differences in pain processing and outcomes. Some researchers have reported the associations between the development of persistent pain, sleep disorders and reduced physical activity. Taken together, these symptoms may lead to disability and worsened quality of life. Due to its benefits, the American Cancer Society recommends to begin as soon as possible from the diagnosis of cancer, physical activity. Aim of this prospective observational study is to evaluate the effects of motor and/or sports activity on the intensity of chronic pain and in symptoms of sleep disorders, caused by post-mastectomy chronic pain. of life of women underwent mastectomy

DETAILED DESCRIPTION:
Chronicization of pain is frequently occurring after surgery, thus leading often to functional limitations and psychological disorders, with a negative impact on quality of life.

Chronic post-surgical pain (CPSP) was first defined as "pain that develops after surgical intervention and lasts at least 2 months; other causes of pain have to be excluded, in particular, pain from a condition existing before the surgery". An updated definition of CPSP, was later proposed as "pain persisting at least three months after surgery, that was not present before surgery, or that had different characteristics or increased intensity from preoperative pain, localized to the surgical site or a referred area, and other possible causes of the pain were excluded (e.g., cancer recurrence, infection)".

Chronic pain following mastectomy, referred to at that time as intercostobrachial nerve entrapment syndrome, was first identified in a case series of patients who underwent mastectomy in the 1970s. This condition is now referred to as post-mastectomy pain syndrome (PMPS). The International Association for the Study of Pain (IASP) defines PMPS as persistent, neuropathic pain that develops soon after mastectomy or lumpectomy located in the anterior surface of the chest axilla, shoulder, or upper half of the arm.

The etiology of persistent pain after mastectomy is still unclear, because of its possible multifactoriality with a partial neuropathic origin. While surgical factors, including axillary lymph node dissection, and reconstruction, have been postulated to serve as important risk factors for chronic pain, many studies do not fully support this association. Adjuvant treatment, such as radiation, chemotherapy, and hormone therapy, has also been occasionally associated with persistent pain consequent to mastectomy.

Psychosocial factors such as anxiety, catastrophizing and sleep disorders are being revealed as crucial contributors to individual differences in pain processing and outcomes. There is substantial evidence supporting the association between chronic pain and sleep, as constant pain affects wakefulness and, consequently, sleep quality. Hence, there is a close relationship between chronic pain and insomnia, and sustained sleep restriction further diminishes emotional and physical well-being, leading to depression, chronic fatigue and anxiety in many patients.

Sleep disturbances have been found to both contribute to and result from immune-neuro-endocrine disorders, which are also associated with the presence of chronic pain in general.

Sleep disturbances encompass both sleep quality and disorders. Sleep quality refers to a multifactorial process encompassing both sleep duration and depth. Sleep disorders are conditions that involve both subjective and objective symptoms, such as insomnia disorders, sleep-related breathing disorders, central disorders of hypersomnolence, circadian rhythm sleep-wake disorders, sleep-related movement disorders, parasomnias, and other sleep disorders.

Humans physiological circadian rhythms is closely associated with sleep quality. The hormones cortisol and melatonin and core body temperature show notable circadian rhythms. Core body temperature decreases at night and increases during daytime. Cortisol and melatonin are counter-regulatory hormones; melatonin levels increase at night, when cortisol levels decrease to their lowest point, and cortisol levels increase to their highest point in the morning, when melatonin levels decrease to their lowest. Abnormal melatonin and cortisol rhythms can cause sleep problems.

Cortisol, a prominent hormone in circadian rhythms, reacts rapidly to exercise, stimulating the sympathetic nervous system as its concentration rapidly increases. Kanaley et al. reported that evening exercise significantly increased cortisol concentrations compared to morning exercise. Additionally, cortisol concentration significantly increases after moderate-intensity exercise compared with low-intensity exercise.

Current evidence indicates that sleep disorders may contribute to the growing health burden in modern societies. Insufficient and poor-quality sleep represent high-risk factors for health outcomes such as cardiovascular disease, cognitive impairment, and metabolic dysfunction; poor sleep has also been associated with risk-taking behavior, accidents, increased mortality rates, and diminished quality of life.

It is well documented that physical activity can improve sleep quality in a variety of ways, increasing the production of melatonin, a hormone that regulates sleep-wake cycles, moreover, several studies suggest that physical activity improves sleep disorders by a modulation of cortisol level and an increase of melatonin levels. Cortisol reacts rapidly to exercise, stimulating the sympathetic nervous system as its concentration rapidly increases. Some studies report that evening exercise significantly increased cortisol concentrations compared to morning exercise. Additionally, cortisol concentration significantly increases after moderate-intensity exercise compared with low-intensity exercise.

As a result, physical activity can assist in falling asleep faster and sleeping better. Second, physical activity reduces stress, which is a typical impediment to falling and staying asleep. Third, physical activity improves mood, leading to increased enthusiasm for physical exercise and a positive feedback loop. It was shown that active people had higher levels of positive affect and tranquility during exercise and lower levels of negative affect and tiredness. Finally, physical activity helps to regulate body temperature, which is necessary for falling asleep, as an increase in body temperature during physical activity aids the eventual drop 30-90 minutes post-exercises, facilitating easier sleepiness.

On the light of the above considerations, the aim of this study was to evaluate the effects of physical activity on the intensity and interference of chronic pain in daily activities and the effect on sleep disturbance in patient underwent mastectomy.

Study population: women underwent unilateral or bilateral mastectomy due to resection of stage II and III breast cancer not followed by breast reconstruction aged 18 years or older who have not received chemotherapy or radiation. Pain assessment: Pain assessment is a multidimensional process, which must take into account all the components of suffering, both physically, psychologically and socially. The assessment of pain and motor activity of each participant in the study will be carried out 3 and 6 months after surgery. Pain will be assessed by administration of Numerical Rating Scale (NRS) questionnaire. For the evaluation of sleep disorders, will be administered the Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI). All the evaluation will be performed 3 and 6 months after surgery. The IPAQ (International Physical Activity Questionnaire) questionnaire measures the type and amount of physical activity that is normally done.

The questions refer to the activity carried out in the last 7 days. It will be administered at 3 and 6 months after surgery.The expected duration of the study can be considered to be approximately 12 months. At the same timepoints (12 and 24 weeks after surgery) hematic biomarkers correlated to pain, and sleep disorders will be measured together with routine blood parameters. Specifically, the following biomarkers will be evaluated: cortisol, adrenocorticotropic hormone (ACTH) and melatonin.

ELIGIBILITY:
Inclusion Criteria: women aging over 18 years with a prior diagnosis of Phase II or III breast cancer who had undergone mastectomy for cancer removal 3 months earlier. -

Exclusion Criteria:

* medical history of other types of cancer;
* disease related to the immune system (e.g. multiple sclerosis, HIV, lupus);
* recent symptoms of illness (cough, fever);
* no antinflammatory or antidepressive or anxiolitic drugs assumption during the first six months after surgery
* waiting breast reconstruction;
* not chemotherapy or radiation during the first six months after surgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aging over 18 yearsunderwent unilateral or bilateral mastectomy due to resection of stage II and III breast cancer.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Effects of motor and/or sports activity on the intensity of chronic pain in women underwent mastectomy. | Evaluation performed three and six months after surgery
  Pain intensity self-measured using the Numerical Rating Scale (NRS). NRS is a 0-11 point-scale where the end points are the extremes of no pain (point 0) and worst pain as bad as it could be (point 10)
Effects of motor and/or sports activity on sleep disorders in women underwent mastectomy suffering by chronic pain. | Evaluation performed three and six months after surgery
  Pittsburgh Sleep Quality Index (PSQI) was used to evaluate the quality of sleep.
  The PSQI is a self-report inventory assessing sleep duration, latency, and overall sleep quality over 1 month time interval. Each item is weighted on a 0-3 interval scale. A score of 0 indicates no difficulty, while a score of 3, indicates severe difficulty. The global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores indicate an healthier sleep quality. A score ≤ 5 generally reflects a good sleep quality while a score > 5 reflects a bad sleep qualityInsomnia Severity Index (ISI) The ISI is a self-rated instrument with seven items that assess insomnia's nature, severity, and impact, rated on a 5-point [0 (no problem) - 4 (very severe problem)]. Insomnia is graded as absent (score 0-7), mild (score 8-14), moderate (score15-21), and severe (score 22-28)

SECONDARY OUTCOMES:
Evaluation of biomarker associated to pain intensity and sleep disorders | Evaluation performed three and six months after surgery]
  Biomarkers correlated to pain intensity and sleep disorders, were evaluated in serum. Analysis was performed in blood aliquot withdrawn during the routine analysis. The following biomarkers were considered: ACTH (pg/mL) and melatonin (pg/mL). All the measures were performed by ELISA according to the manufacturer protocol.
Evaluation of serum cortisol | Evaluation performed three and six months after surgery
  Serum cortisol (ng/mL) was evaluated by ELISA analysis, according to the manufaturer protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Gioacchino Calapai, Messina, Italy, Italy

REFERENCES:
- [Background] Calapai M, Esposito E, Puzzo L, Vecchio DA, Blandino R, Bova G, Quattrone D, Mannucci C, Ammendolia I, Mondello C, Gangemi S, Calapai G, Cardia L. Post-Mastectomy Pain: An Updated Overview on Risk Factors, Predictors, and Markers. Life (Basel). 2021 Sep 29;11(10):1026. doi: 10.3390/life11101026. PMID 34685397
- [Background] Magnan RE, Kwan BM, Bryan AD. Effects of current physical activity on affective response to exercise: physical and social-cognitive mechanisms. Psychol Health. 2013;28(4):418-33. doi: 10.1080/08870446.2012.733704. Epub 2012 Oct 23. PMID 23088712
- [Background] Ambrose KR, Golightly YM. Physical exercise as non-pharmacological treatment of chronic pain: Why and when. Best Pract Res Clin Rheumatol. 2015 Feb;29(1):120-30. doi: 10.1016/j.berh.2015.04.022. Epub 2015 May 23. PMID 26267006
- [Derived] Calapai M, Puzzo L, Bova G, Vecchio DA, Blandino R, Barbagallo A, Ammendolia I, Cardia L, Firenzuoli F, Calapai F, Curro M, Ficarra G, Esposito E, Trimarchi F, Di Mauro D, Calapai G, Mannucci C. Post-mastectomy pain syndrome and sleep disorders: effects of physical activity. Front Sports Act Living. 2025 Nov 20;7:1579635. doi: 10.3389/fspor.2025.1579635. eCollection 2025. PMID 41357821
- See also: There are no website that provide information that is directly related to the study protocol — http://www.unime.it